CLINICAL TRIAL: NCT06181643
Title: Innovating CBT-I for Cancer Survivors: An Optimization Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel L Hall, PhD, Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-681
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cancer Survivorship; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Survivorship Sleep Program with Individual Delivery + No Booster Sessions (Experimental): 4 weekly SSP sessions delivered to individual participants (session durations approximately 45 min/session). No booster sessions.
  Interventions: Behavioral: Survivorship Sleep Program with Individual Delivery + No Booster Sessions
- Group 2: Survivorship Sleep Program with Group Delivery + No Booster Sessions (Experimental): 4 weekly SSP sessions delivered to groups of participants (session durations approximately 90 min/session). No booster sessions.
  Interventions: Behavioral: Survivorship Sleep Program with Group Delivery + No Booster Sessions
- Group 3: Survivorship Sleep Program with Individual Delivery + 3 Booster Sessions (Experimental): 4 weekly SSP sessions delivered to individual participants (session durations approximately 45 min/session), followed by 3 monthly booster sessions.
  Interventions: Behavioral: Survivorship Sleep Program with Individual Delivery + 3 Booster Sessions
- Group 4: Survivorship Sleep Program with Group Delivery + 3 Booster Sessions (Experimental): 4 weekly SSP sessions delivered to groups of participants (session durations approximately 90 min/session), followed by 3 monthly booster sessions.
  Interventions: Behavioral: Survivorship Sleep Program with Group Delivery + 3 Booster Sessions

INTERVENTIONS:
Behavioral: Survivorship Sleep Program with Individual Delivery + No Booster Sessions — 4 weekly SSP sessions delivered to individual participants (session durations approximately 45 min/session). No booster sessions.
  Arms: Group 1: Survivorship Sleep Program with Individual Delivery + No Booster Sessions
Behavioral: Survivorship Sleep Program with Group Delivery + No Booster Sessions — 4 weekly SSP sessions delivered to groups of participants (session durations approximately 90 min/session). No booster sessions.
  Arms: Group 2: Survivorship Sleep Program with Group Delivery + No Booster Sessions
Behavioral: Survivorship Sleep Program with Individual Delivery + 3 Booster Sessions — 4 weekly SSP sessions delivered to individual participants (session durations approximately 45 min/session). 3 monthly booster sessions.
  Arms: Group 3: Survivorship Sleep Program with Individual Delivery + 3 Booster Sessions
Behavioral: Survivorship Sleep Program with Group Delivery + 3 Booster Sessions — 4 weekly SSP sessions delivered to groups of participants (session durations approximately 90 min/session). 3 monthly booster sessions.
  Arms: Group 4: Survivorship Sleep Program with Group Delivery + 3 Booster Sessions

SUMMARY:
The overall goal of this project is to conduct a factorial, randomized controlled trial to optimize synchronous, virtual delivery of CBT-I for cancer survivors. The proposed project will yield multiple deliverables to innovate cancer survivorship care, chiefly an optimized, scalable, virtually-delivered intervention that addresses chronic insomnia, one of the most deleterious concerns among the growing demographic of cancer survivors in the U.S. Findings will inform future considerations for delivering CBT-I to cancer survivors.

DETAILED DESCRIPTION:
Insomnia is a significant issue in 30-50% of cancer survivors. Our pilot randomized controlled trial of synchronous, virtual cognitive behavioral therapy for insomnia (CBT-I) for cancer survivors suggested that a group format or booster sessions may optimize effects on insomnia and daytime functioning. The goal of this project is to conduct a factorial, randomized controlled trial to optimize synchronous, virtual delivery of CBT-I for cancer survivors. We will conduct a 2×2 factorial trial (N=80) to evaluate the optimal combination of two intervention design components: delivery (individual vs. group) and booster sessions (0 vs 3). The primary outcome is change in insomnia severity (insomnia severity index) from T0 (week 0) to T2 (week 8). The secondary outcomes are acute (T0-T1, week 4) and sustained (T0-T3, week 16) changes in insomnia severity, emotional distress, work-related functioning, use of sleep medications, and subjective and objective sleep metrics (measured with sleep diaries and Fitbit). Exploratory aim 1 is to characterize study participation and sleep outcomes among cancer survivors with insomnia. Exploratory aim 2 is to characterize the acceptability of design components using Likert ratings (very low=1 to very high=5, benchmarks=4 or higher) and exit interviews with open-ended responses with probes. This project will yield multiple deliverables to innovate cancer survivorship care, chiefly an optimized, scalable, virtually delivered intervention that addresses chronic insomnia, one of the most deleterious concerns among the among the steadily increasing number of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* History of nonmetastatic, localized, or regional solid or blood malignancy(ies)
* Completion of primary cancer treatment (radiation, surgery, and/or chemotherapy). Use of hormonal, maintenance, oral, and immunotherapies is permitted.
* Chronic insomnia (DSM-5 criteria)
* 18 years of age or older

Exclusion Criteria:

* Self-reported inability to speak and write in English
* Undertreated noninsomnia sleep disorder (e.g., sleep apnea)
* Undertreated epilepsy, undertreated serious mental illness, undertreated suicidality, and/or psychiatric hospitalization in the past year
* Unwilling or unable to discontinue night shift work

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) total score | T0 (Baseline) to T2 (week 8)
  Changes in insomnia severity will be assessed using the validated Insomnia Severity Index (ISI). Scores of 15 or higher on the ISI indicate clinically significant insomnia, and reductions of >8 points are considered clinically meaningful. Changes from T0-T2 are the primary outcome. Acute (T0-T1; post-SSP) and 3-month (T0-T3; 3 Month Surveillance/Booster 3) changes will be examined as secondary outcomes.

SECONDARY OUTCOMES:
Emotional distress: PROMIS Anxiety Symptoms | T0 (week 0) to T3 (week 16)
  PROMIS anxiety short form. Acute (T0-T1; week 4) and 3-month (T0-T3; week 16) changes will be examined as secondary outcomes.
Emotional distress: PROMIS Depression Symptoms | T0 (week 0) to T3 (week 16)
  PROMIS depression short form. Acute (T0-T1; week 4) and T0-T3 (week 16) changes will be examined as secondary outcomes.
Daytime fatigue: PROMIS Fatigue | T0 (week 0) to T3 (week 16)
  PROMIS fatigue short form. Acute (T0-T1; week 4) and T0-T3 (week 16) changes will be examined as secondary outcomes.
Work-related functioning | T0 (week 0) to T3 (week 16)
  Work-related functioning will be measured using the six-item Work Productivity and Activity Impairment: General Health (WPAI:GH), which includes scores for absenteeism, presenteeism, and total work impairment. Acute (T0-T1; week 4) and T0-T3 (week 16) changes will be examined as secondary outcomes.
Use of sleep aid medications | T0 (week 0) to T3 (week 16)
  Use of sleep aid medications (frequency, dose) will be evaluated via self-report surveys and electronic medical records (when possible). Acute (T0-T1; week 4) and T0-T3 (week 16) changes will be examined as secondary outcomes.
Sleep diaries and actigraphy | T0 (week 0) to T3 (week 16)
  Sleep diaries and actigraphy will be collected during SSP Sessions 1-4 and for 7 days at each timepoint (T0-T3) to derive sleep efficiency, sleep onset latency, and wake after sleep onset. Discrepancy scores between subjective and objective sleep metrics (e.g., sleep onset latency) will be examined. Acute (T0-T1; week 4) and T0-T3 (week 16) changes will be examined as secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hall, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States